CLINICAL TRIAL: NCT03307512
Title: Samba-AC: A Randomized, Open-Label, Cross-Over Study to Investigate the PK and PD Profiles of Dance 501 (Human Insulin Inhalation Solution and Inhaler) in Healthy Subjects and Non-Diabetic Subjects With Mild to Moderate Asthma or COPD
Brief Title: PK and PD Profile of Dance 501 in Healthy, Non-diabetic Subjects With Mild to Moderate Asthma or COPD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination due to incomplete enrollment; planned data analysis not performed
Sponsor: Dance Biopharm Inc. (Industry)
Collaborators: WCCT Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Samba-AC
Record Dates: First submitted 2017-10-02; First posted 2017-10-11 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Safety and Tolerability
Keywords: inhaled insulin; asthma; COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, cross-over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dance 501 (Experimental): Dance 501(Human Insulin Inhalation Solution and Inhaler) will be administered by inhalation
  Interventions: Drug: inhaled human insulin
- Insulin Lispro (Active Comparator): Insulin Lispro (Humalog®) will be administered by subcutaneous injection
  Interventions: Drug: Insulin Lispro (Humalog U-100)

INTERVENTIONS:
Drug: inhaled human insulin — Dance 501 (Human Insulin Inhalation Solution and Inhaler) will be administered by inhalation
  Other Names: Dance 501
  Arms: Dance 501
Drug: Insulin Lispro (Humalog U-100) — Insulin Lispro (Humalog U-100) will be administered by subcutaneous injection
  Other Names: Lispro
  Arms: Insulin Lispro

SUMMARY:
This will be a randomized, open-label, active-controlled, single dose crossover study with either three or four treatment periods. Investigational treatment is with Dance 501 Human Insulin Inhalation Solution (Dance 501) and the comparator is Insulin Lispro (Humalog®).

Target population will be Non-Diabetic individuals with mild to moderate asthma or chronic obstructive pulmonary disease (COPD) and non-diabetic individuals without underlying lung disease (healthy subjects).

DETAILED DESCRIPTION:
The PK and PD profile of Dance 501 (Human Insulin Inhalation Solution and Inhaler) will be compared to subcutaneous injection of insulin lispro.

ELIGIBILITY:
Inclusion Criteria:

* non-diabetic subjects with asthma, or COPD. Non-smokers or smokers quit at least 6 months prior to enrollment. BMI <= 35 kg/m2. Fasting blood glucose <= 125 mg/dL.

Exclusion Criteria:

* pulmonary disorder other than asthma or COPD. Upper respiratory within previous 4 weeks. Significant exacerbation of asthma or COPD symptoms. Hospitalization for asthma or COPD within previous 3 months. Clinically significant medical condition. Current medications interfering with glucose metabolism.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Area under the insulin curve (AUC) | 10 hours
  Area under the insulin curve (AUC)
Area under the glucose infusion rate curve (GIR) | 10 hours
  Area under the glucose infusion rate curve (GIR)

SECONDARY OUTCOMES:
Area under the insulin curve following inhalation of salbutamol | 10 hours
  Area under the insulin curve following inhalation of salbutamol in subjects with asthma

CONTACTS AND LOCATIONS:
Overall Officials: Timothy S Bailey, MD, Principal Investigator — AMCR
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No